CLINICAL TRIAL: NCT00000728
Title: Phase I Trial of the Combination of Zidovudine and Recombinant Interleukin-2 in Patients With Persistent Generalized Lymphadenopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 024; 11000 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Immune Tolerance; Interleukin-2; Drug Therapy, Combination; AIDS-Related Complex; Zidovudine; CD4-Positive T-Lymphocytes
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Zidovudine; aldesleukin

INTERVENTIONS:
Drug: Zidovudine
Drug: Aldesleukin

SUMMARY:
To evaluate the short-term effects of administering zidovudine ( AZT ) at the same time with increasing doses of aldesleukin ( interleukin-2; IL-2 ) in patients with persistent generalized lymphadenopathy syndrome ( PGL ). The effects to be studied include safety or toxicity, how quickly the drugs are used in the body, effects on the immune system, effects on HIV, concentrations in body fluids, and how quickly the drugs are cleared by the kidneys. The trial will establish the maximum tolerated dose ( MTD ) and will be a pilot study to determine the dose that has the greatest effect in the immune system.

AZT has been shown to be effective in HIV-related disease. IL-2 has been shown to increase immune responses and correct immune problems caused by HIV in the test tube. IL-2 has also been effective in treating Kaposi's sarcoma in a number of patients. Because of the clinical activities of these two drugs and because their toxicities and mechanisms of action do not overlap, it may be beneficial to combine the two drugs with their antiviral and immune stimulatory effects.

DETAILED DESCRIPTION:
AZT has been shown to be effective in HIV-related disease. IL-2 has been shown to increase immune responses and correct immune problems caused by HIV in the test tube. IL-2 has also been effective in treating Kaposi's sarcoma in a number of patients. Because of the clinical activities of these two drugs and because their toxicities and mechanisms of action do not overlap, it may be beneficial to combine the two drugs with their antiviral and immune stimulatory effects.

Patients enter the study in staggered groups of five. All patients receive AZT orally every 4 hours for 12 weeks. At the end of 8 weeks, the first group of five patients receive the lowest dosage of IL-2 on a daily basis while still receiving AZT. Toxicity and immunologic effects are measured at the beginning of AZT therapy and then every 2 weeks. Each succeeding group of five patients receives a higher dose of IL-2, while receiving AZT, until the MTD is reached. Those patients who have shown no toxicity as well as improved immune function while taking both drugs receive a 4-week follow-up course of IL-2 5 weeks after stopping AZT. In addition, five patients who have completed the AZT / IL-2 combined treatment without significant toxicity are re-treated with 12 weeks of AZT alone starting 8 weeks after completing the initial combined AZT / IL-2 portion of treatment. Another five patients will be re-treated with 12 weeks of full dose of AZT alone, followed by 8 weeks of half-dose AZT alone starting 8 weeks after completing the initial combined AZT / IL-2 treatment. Patients receive ibuprofen for fever and chills, and those who reach their MTD continue to receive that dose in combination with AZT for 4 weeks. If excess toxicity is observed on all doses of IL-2, the study will be discontinued.

ELIGIBILITY:
Inclusion Criteria

* Detectable HIV nucleic acid in patient peripheral blood mononuclear leukocytes (PBML's) by the gene amplification technique. A positive antibody to HIV confirmed by any federally licensed ELISA test kit.

Concurrent Medication:

Allowed:

* Medications without which there might be significant risk, such as seizures, loss of diabetic control or respiratory embarrassment.
* Necessary topical agents including topical acyclovir.
* Diuretics for significant fluid retention only.

Concurrent Treatment:

Allowed:

* Blood transfusions for anemia if hematocrit falls below 25 percent.

Exclusion Criteria

* Active drug or alcohol abuse.

Co-existing Condition:

Patients with the following will be excluded:

* Grade 1 impairment on two or more items in the ACTG Micro Neuro AIDS assessment.
* Concurrent neoplasms other than basal cell carcinoma of the skin or in situ carcinoma of the cervix.
* Major organ allograft.
* Significant cardiac disease or central nervous system lesions.
* Patients with hemophilia should be evaluated and treated under the hemophilia protocol.

Concurrent Medication:

Excluded:

* Inderal or vasoactive hypertensive medication.
* Non-essential medications including pain medications.

Excluded are:

* Patients with an opportunistic infection or malignancy fulfilling the definition of AIDS.

Patients with AIDS related complex, defined as:

* 1. Weight loss in excess of 15 lbs. or 10 percent of body weight noted in a 2-year period prior to entry into the study. 2. Temperature greater than 38.5 degrees C with or without night sweats, persisting for more than 14 consecutive days or more than 15 days in a 30-day interval during a 2-year period prior to entry into the study. 3. Diarrhea defined as = or > 3 liquid stools per day, persisting for more than 30 days during a 2-year period prior to entry into the study without a definable cause. 4. Herpes zoster during the past 2 years. 5. Oral candidiasis or biopsy-proven hairy leukoplakia during the last 2 years. 6. Active substance abuse.

Prior Medication:

Excluded:

* Zidovudine (AZT).
* Excluded within 30 days of study entry:
* Antiretroviral agents.
* Biologic response modifiers.
* Corticosteroids.
* Excluded within 60 days of study entry:
* Ribavirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Study Completion 1990-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merigan TC, Study Chair
Locations (1):
- Stanford Univ School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Schwartz DH, Skowron G, Merigan TC. Safety and effects of interleukin-2 plus zidovudine in asymptomatic individuals infected with human immunodeficiency virus. J Acquir Immune Defic Syndr (1988). 1991;4(1):11-23. PMID 1670586